CLINICAL TRIAL: NCT01483248
Title: Phase 1/2 Study of Human Menstrual Blood-derived Mesenchymal Stem Cells Transplantation for the Evaluation of the Efficacy and Safety in Patients With Liver Cirrhosis
Brief Title: Human Menstrual Blood-derived Mesenchymal Stem Cells for Patients With Liver Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: S-Evans Biosciences Co., Ltd. (Industry)
Collaborators: Zhejiang University (Other); Zhejiang General Hospital of Armed Police (Other); Zhenjiang First People's Hospital (Other); Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEB-1115-LC
Record Dates: First submitted 2011-11-23; First posted 2011-12-01 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Liver Cirrhosis; Fibrosis; Liver Disease; Digestive System Disease
Keywords: Menstrual blood; Mesenchymal stem cell; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Liver Diseases; Digestive System Diseases | interventions — Interferons; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Conventional therapy plus MenSCs treatment
  Interventions: Biological: conventional therapy plus MenSC transplantation
- No intervention (Active Comparator): Conventional therapy plus placebo treatment:
  Oral or intravenous administration
  Interventions: Drug: Conventional therapy plus placebo treatment

INTERVENTIONS:
Biological: conventional therapy plus MenSC transplantation — patients will receive conventional treatment,such as antiviral drugs, lowering aminotransferase and jaundice medicine.
  MenSCs transplantation: taken i.v., twice per week, at a dose of 1*10E6 MSC/kg body for 2 weeks.
  Other Names: Interferon; Bifendatatum; Ursodeoxycholic Acid; Menstrual blood-derived stem cells(MenSCs)
  Arms: Intervention
Drug: Conventional therapy plus placebo treatment — 25 of the enrolled patients were assigned to receive comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine.
  Other Names: Interferon; Bifendatatum; Ursodeoxycholic Acid
  Arms: No intervention

SUMMARY:
Orthotopic liver transplantation (OLT) is currently the most effective method for end-stage liver diseases. However, the critical shortage of donor organs, high cost, and the problem of immune rejection limit its clinical application, and even some patients on the waiting list will never survive to receive a matched liver. Stem cell transplantation instead of conventional medical therapy or orthotopic liver transplantation will be a promising alternate approach to regenerate damaged hepatic mass. Adult mesenchymal stem cells (MSCs) are generally thought of as an autologous source of regenerative cells in previous studies.In this study, the safety and efficacy of menstrual blood-derived stem cells transplantation for patients with liver cirrhosis will be evaluated.

DETAILED DESCRIPTION:
The purpose of this study is to show whether menstrual blood-derived stem cells can improve the disease conditions in patients with liver cirrhosis.

One of two treatment arms will be assigned to the patients. One group will receive 2 weeks of conventional therapy plus MenSCs treatment; The other group will receive 2 weeks of conventional therapy plus placebo treatment.

MenSCs will be cultured and collected in a GMP lab. Patients were strictly monitored after the cells injection via i.v.. Patients are followed up at intervals up to at least 2 years.Clinical parameters such as ascites volume,serum alanine aminotransferase,total bilirubin,prothrombin time,albumin,MELD score,and Child-Pugh score will be evaluated at each timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged 20 to 50years
* Liver cirrhosis
* Negative pregnancy test

Exclusion Criteria:

* Pregnant or lactating women
* Malignancies
* Sepsis
* Vital organs failure
* Severe bacteria infection
* Vascular thromboses in the portal or hepatic veins

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 48 weeks

SECONDARY OUTCOMES:
Liver function improvement | 48 weeks
Complications | 48 weeks
  such as fever,anaphylaxis,cough,chest distress,and dyspnea,et al.
The improvement of ascites after 12-week treatment | 48 weeks
Child-Pugh score | 48 weeks
MELD score | 48 weeks
SF36-quality of life | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Xiang, Professor, Principal Investigator — S-Evans Biosciences Co., Ltd.
Locations (1):
- the First Affiliated Hospital of Zhejiang University-IRB, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Houlihan DD, Hopkins LJ, Suresh SX, Armstrong MJ, Newsome PN. Autologous bone marrow mesenchymal stem cell transplantation in liver failure patients caused by hepatitis B: short-term and long-term outcomes. Hepatology. 2011 Nov;54(5):1891-2; author reply 1892. doi: 10.1002/hep.24722. No abstract available. PMID 21987440
- [Background] Peng L, Xie DY, Lin BL, Liu J, Zhu HP, Xie C, Zheng YB, Gao ZL. Autologous bone marrow mesenchymal stem cell transplantation in liver failure patients caused by hepatitis B: short-term and long-term outcomes. Hepatology. 2011 Sep 2;54(3):820-8. doi: 10.1002/hep.24434. Epub 2011 Jul 14. PMID 21608000
- [Background] Forbes SJ, Newsome PN. New horizons for stem cell therapy in liver disease. J Hepatol. 2012 Feb;56(2):496-9. doi: 10.1016/j.jhep.2011.06.022. Epub 2011 Jul 26. PMID 21798218
- [Background] Nikeghbalian S, Pournasr B, Aghdami N, Rasekhi A, Geramizadeh B, Hosseini Asl SM, Ramzi M, Kakaei F, Namiri M, Malekzadeh R, Vosough Dizaj A, Malek-Hosseini SA, Baharvand H. Autologous transplantation of bone marrow-derived mononuclear and CD133(+) cells in patients with decompensated cirrhosis. Arch Iran Med. 2011 Jan;14(1):12-7. PMID 21194255
- [Background] Zhang D, Jiang M, Miao D. Transplanted human amniotic membrane-derived mesenchymal stem cells ameliorate carbon tetrachloride-induced liver cirrhosis in mouse. PLoS One. 2011 Feb 4;6(2):e16789. doi: 10.1371/journal.pone.0016789. PMID 21326862
- See also: North American Indian childhood cirrhosis — http://ghr.nlm.nih.gov/
- See also: Cirrhosis — http://www.nlm.nih.gov/medlineplus/
- See also: Related Info — http://www.fda.gov/